CLINICAL TRIAL: NCT05934084
Title: Lifestyles Implemented-Survivorship Care Plan In Lymphoma Survivors: A Randomized Non-pharmacological Clinical Trial By The Fondazione Italiana Linfomi (FIL)
Brief Title: Lifestyles Implemented-Survivorship Care Plan In Lymphoma Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FIL_Lymphoma-SCP
Record Dates: First submitted 2023-06-13; First posted 2023-07-06 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Classical Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma (DLBCL); Primary Mediastinal Large B-cell Lymphoma (PMBCL)
Keywords: Survivorship Care Plan; Lifestyles implemented-Survivorship Care Plan; Quality of Life; Lymphoma Survivors; Nutritional plan; Physical activity
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Motor Activity

STUDY DESIGN:
Intervention Model Description: It's a longitudinal study with two time-points (6 months and 12 months) after baseline (time 0) and the data will be evaluated by means of ANOVA for repeated measures, considering as baseline the global QoL of 75.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (C) (No Intervention): Patients in the control arm will not receive any Survivorship Care Plan (SCP) or intervention and will be followed-up according to the best clinical practice, with questionnaires self-administration at 6 and 12 months from randomization.
- Experimental Arm (E) (Experimental): Patients in the experimental arm will follow the planned intervention (Survivorship Care Plan (SCP), nutritional plan, physical activity indication) for 6 months.
  Interventions: Behavioral: Lifestyles Implemented-Survivorship Care Plan (LS-SCP)

INTERVENTIONS:
Behavioral: Lifestyles Implemented-Survivorship Care Plan (LS-SCP) — Patients in the experimental arm will follow the planned intervention (Survivorship Care Plan (SCP), nutritional plan, physical activity) for 6 months. A bi-monthly automatic call to assess the compliance at the experimental arm (LS-SCP, Lifestyles implemented-Survivorship Care Plan) will be performed.
  Arms: Experimental Arm (E)

SUMMARY:
This is a prospective randomized open-label, multicenter, 2-arm study to assess the role of healthy LifeStyle implemented Survivorship Care Plan (LS-SCP) in modifying the Quality of Life (QoL) in a population of long-term lymphoma survivors (in remission for a minimum 3 years since the last treatment and a maximum of 10 years).

DETAILED DESCRIPTION:
All patients will be assessed by validated questionnaires [EORTC QLQ-C30 (Quality of Life Questionnaire), SF12 (12-item Short Form Survey), MEDI-LITE (Mediterranean Literature questionnaire), CFSS (Chronic Fatigue Syndrome Self assessment), FAS (Fatigue Assessment Scale), Hospital Anxiety and Depression Scale (HAD-S)] and clinical assessment performed at baseline, at 6 and 12 months from the randomization. Patients in the experimental arm will follow the planned intervention (Survivorship Care Plan (SCP), nutritional plan, physical activity) for 6 months. A bi-monthly automatic call to assess the compliance at the experimental arm (Lifestyles implemented-Survivorship Care Plan (LS-SCP)) will be performed. Patients in the control arm will not receive any Survivorship Care Plan (SCP) or intervention and will be followed-up according to the best clinical practice, with questionnaires self-administration at 6 and 12 months from randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 at initial treatment;
* Diagnosis of classical Hodgkin lymphoma (cHL), Diffuse Large B-cell lymphoma (DLBCL) or Primary mediastinal large B-cell lymphoma (PMBCL);
* Patients in Complete Remission (CR) after first-line therapy [ABVD (doxorubicin, bleomycin, vinblastine, dacarbazine) or BEACOPP (bleomycin, etoposide, doxorubicin , cyclophosphamide, vincristine, procarbazine and prednisone) or ABVD-BEACOPP Pet-2 guided treatment for cHL; R-CHOP (rituximab-cyclophosphamide, doxorubicin, vincristine and prednisone) for DLBCL; R-CHOP or R-DA-EPOCH (rituximab- Dose Adapted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin) for PMBCL);
* Patients in remission for a minimum 3 years since the last treatment and a maximum of 10 years;
* Cumulative doxorubicin/ adriamycin dose received of at least 200 mg/mq (4 cycles of chemotherapy);
* Availability echocardiogram (ECG) and 2D-STE-echocardiography (Two-dimensional speckle strain echocardiography) performed no later than three months prior to enrollment;
* Signature of a written informed consent form indicating that the patient understands the purpose of and procedures required for the study and is willing to participate voluntarily in the study.

Exclusion Criteria:

* Diagnosis of secondary cancer at baseline, except non-melanoma skin cancers and adequately treated cone-biopsied in situ carcinoma of the cervix;
* Second line chemotherapy of stem cell transplant;
* Not able to perform physical activity;
* Grade >/=3 neuropathy;
* Vertebral fractures or stenosis of the vertebral canal; other bone fracture;
* Cardiovascular disease: arrhythmia >/= grade 2, hypertension >/ grade 2, left ventricular dysfunction >/= grade 2 pericardial disease/effusion any grade, myocarditis any grade, pulmonary hypertension any grade, restrictive cardiomyopathy any grade valvular hearth disease >/= grade 2, right ventricular dysfunction >/= grade 2;
* Venous thromboembolism or arterial thrombosis during last 6 months;
* Hemorrhage/ bleeding >/= grade 2 during last 6 months;
* Chronic lymphedema (arms and/ or limbs);
* Rheumatic disease or inflammatory bowel disease in systemic treatment;
* Any pleural effusion;
* If female, the patient is pregnant;
* Unwilling to comply to all required visits and procedures for the duration of study participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 552 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Global quality of life | From study start up to 30 months
  The endpoint will be assessed by the European Organisation For Research And Treatment Of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) that will be submitted to patients.
  The EORTC QLQ-C30 consists of 30 items including five functioning scales (physical functioning, social functioning, role functioning, emotional functioning and cognitive functioning), nine symptom scales (fatigue, pain, nausea-vomiting, dyspnoea, sleep disturbances, appetite loss, diarrhoea, constipation and financial difficulties), and a global health status or quality of life (QOL) scale. On the 100-point metric, high scores for functioning scales and the global health status, or QOL, scale indicate high HR (health-related) QOL, while high scores on the symptom scales indicate a high symptom burden.

SECONDARY OUTCOMES:
Impact of health on an individual's everyday life | From study start up to 30 months
  The endpoint will be assessed by the 12-Item Short Form Survey (SF-12) which will be submitted to patients. Survey scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Changes in psychosocial well-being | From study start up to 30 months
  The endpoint will be assessed by Hospital Anxiety and Depression Scale (HAD-S) questionnaire which will be submitted to patients. The HAD-S questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Overall survival (OS) | From study start up to 30 months
  Overall survival, the percentage of patients alive of the cohort
Frequencies of chronic fatigue (FAS); | From study start up to 30 months
  The number of times chronic fatigue is recorded in the cohort of patients
Cognitive function | From study start up to 30 months
  The endpoint will be assessed by Cognitive Functioning Self-Assessment Scale (CFSS) questionnaire which will be submitted to patients.
  The Cognitive Functioning Self-Assessment Scale (CFSS) is a questionnaire designed for the self-reporting of cognitive functioning.
  Its 18 items cover cognitive domains such as attention, memory and spatial-temporal orientation. Each item describes an activity of daily life in which these domains are involved. Participants answer each item on a 5-point frequency scale, referring to the past 12 months. The tool provides an overall score, calculated as the mean of the scores on individual items, where higher values indicate a worse self-perception regarding cognitive functioning.
Metabolic outcomes -BMI | From study start up to 30 months
  Body Mass Index (BMI) will be evaluated for every patient. Weight and height will be combined to report BMI in kg/m^2.
Metabolic outcomes - diabetes | From study start up to 30 months
  Number of patients of the cohort with diabetes
Frequency cardiovascular disease | From study start up to 30 months
  The number of times cardiovascular disease is observed in the cohort of patients
Compliance to screening for secondary cancers and vaccination | From study start up to 30 months
  The number of times patients undergo screening and prevention for secondary cancers
Frequency others comorbidity | From study start up to 30 months
  The number of times others comorbidities are observed in the cohort of patients
Adherence to healthy lifestyles - healthy diet | From study start up to 30 months
  The endpoint will be assessed by MEDI-LITE (Mediterranean Literature) questionnaire that will be submitted to patients. Adherence to the Mediterranean diet assessed through the Medi-Lite score was found to be associated with abdominal obesity. The final score, obtained by summing these values, varies from 0 (low adherence) to 18 (high adherence).
Adherence to healthy lifestyles - Physical Activity | From study start up to 30 months
  The endpoint will be assessed by IPAQ (International Physical Activity Questionnaire) that will be submitted to patients. This questionnaire measures the type and amount of physical activity the patient normally does. The questions refer to activity during the past 7 days at work, getting from place to place, and during leisure time. For the purpose of the questionnaire: one minute per week (MET) is what a patient consumes at rest. Therefore, 2 METS is twice what a patient spends at rest. To obtain a continuous variable score from the IPAQ (MET minutes per week), we will consider walking as 3.3 METS, moderate physical activity as 4 METS, and vigorous physical activity as 8 METS.
Measure of hand grip muscle strength | From study start up to 30 months
  This end point will be measured through the use of the hand-grip dynamometer
Frequencies of negative Life-Style factors | From study start up to 30 months
  Number of negative Life-Style factors associated with cardiotoxicity and metabolic syndrome.
Frequency of compliance between planned and effective follow-up via LS-SCP. | From study start up to 30 months
  Number of times the plan prescribed by the LS-SCP is adhered to correctly in the cohort of patients

CONTACTS AND LOCATIONS:
Overall Officials: Carla Minoia, MD, Principal Investigator — Bari, IRCCS Istituto Tumori Giovanni Paolo II - U.O.C Ematologia
Locations (40):
- Italy (40):
  - Ancona - AOU Ospedali Riuniti - Clinica di Ematologia, Ancona, Ancona
  - Aviano - IRCCS Centro di Riferimento Oncologico di Aviano - Divisione di Oncologia e dei Tumori immuto-correlati, Aviano, Aviano
  - Istituto Tumori Bari Giovanni Paolo II, U.O. di Ematologia e Terapia Cellulare, Bari, Bari
  - Ospedale S. Martino - UOC Oncologia, Belluno, Belluno
  - Ospedale "Monsignor Raffaele Dimiccoli" - Ematologia, Barletta
  - Ospedale Centrale di Bolzano - Divisione di Ematologia e T.M.O., Bolzano
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - Ospedale Antonio Perrino - U.O. Ematologia e Trapianti di Midollo, Brindisi
  - PO Sant'Elia ASP Caltanisetta - UOC Ematologia, Caltanissetta
  - Arnas Nuovo Ospedale Garibaldi Nesima - U.O.C. Ematologia, Catania
  - Azienda Ospedaliera Universitaria Policlinico - S. Marco - UOC di Emtologia, Catania
  - Ospedale Generale di zona Valduce - Oncoematologia, Como
  - Azienda Ospedaliera Universitaria Careggi - Unitа funzionale di Ematologia, Florence
  - Ospedale Vito Fazzi - Ematologia, Lecce
  - ASST Ovest Milanese - Legnano - U.O.C. Ematologia Ospedale Civile di Legnano, Legnano
  - AOU G. Martino - U.O.C. Ematologia, Messina
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan
  - IEO Istitito Europeo di Oncologia - Divisione Ematoncologia, Milan
  - Ospedale Maggiore Policlinico - Fondazione IRCCS Ca Granda - Ematologia, Milan
  - Azienda Ospedaliero-Universitaria Policlinico di Modena - U.O. Oncologia, Modena
  - AOU Maggiore della Caritа di Novara - SCDU Ematologia, Novara
  - AOU di Padova - Ematologia, Padua
  - I.R.C.C.S. Istituto Oncologico Veneto - Oncologia 1, Padua
  - Presidio ospedaliero "A. TORTORA" - U.O. Onco-ematologia, Pagani
  - AOU Policlinico Giaccone - Ematologia, Palermo
  - P.O. Spirito Santo di Pescara - UOS Dipartimentale - Centro di diagnosi e Terapia dei linfomi, Pescara
  - Ospedale Guglielmo da Saliceto - U.O.Ematologia, Piacenza
  - AOU Pisana - U.O. Ematologia, Pisa
  - A.O.R. "San Carlo" - U.O. Ematologia, Potenza
  - Azienda Unità Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova - Ematologia, Reggio Emilia
  - Ospedale degli Infermi di Rimini - U.O. di Ematologia, Rimini
  - AO Sant'Andrea - Ematologia, Roma
  - Ospedale S. Eugenio - UOC Ematologia, Roma
  - Policlinico Tor Vergata - Ematologia, Roma
  - Policlinico Universitario Campus Bio-Medico - Ematologia - Trapianto cellule staminali - Medicina Trasfusionale e Terapia cellulare, Roma
  - Istituto Clinico Humanitas - U.O. Ematologia, Rozzano
  - AOU di Sassari - Ematologia, Sassari
  - Nuovo Ospedale Civile di Sassuolo - Day Hospital Oncologico, Sassuolo
  - A.O.U. Citta della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - Ospedale Ca Foncello - S.C di Ematologia, Treviso

IPD SHARING:
Plan to Share IPD: No